CLINICAL TRIAL: NCT00160030
Title: Phase II Study Comparing Radiochemotherapy With the Folfox 4 Regimen Versus Radiochemotherapy With 5FU-Cisplatin (Herskovic Regimen) in First Line Treatment of Patients With Inoperable Esophageal Cancer
Brief Title: Study Comparing Radiochemotherapy With Folfox 4 Regimen or 5FU-Cisplatin in Patients With Inoperable Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_9326
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: FOLFOX 4
- 2 (Active Comparator)
  Interventions: Drug: 5-FU / Cisplatin

INTERVENTIONS:
Drug: FOLFOX 4 — total treatment of six 2-weekly cycles of FOLFOX 4, the first 3 cycles starting on D1, D15 and D29 concomitant with 5 weeks' radiotherapy.
  Arms: 1
Drug: 5-FU / Cisplatin — two cycles of 5-FU / Cisplatin on week 1 and 5 of radiotherapy and two cycles of chemotherapy with 5-FU / Cisplatin on week 8 and 11 (one cycle each three weeks after the end of radiotherapy).
  Arms: 2

SUMMARY:
The primary objectives of this study are to assess the feasibility (completion of full treatment) in both arms and to assess endoscopic complete response rate in both arms.

The secondary objective of this study is to assess the toxicity profile of each arm using the National Cancer Institute-Common Toxicity Criteria (NCI-CTC) scale (V.3).

ELIGIBILITY:
Inclusion Criteria:

Patients with:

* Histologically proven adenocarcinoma, squamous cell or adenosquamous carcinoma of the esophagus
* Inoperable esophageal carcinoma (disease status: any T, N0 or N1, M0 or M1a) or surgical contraindication conditions
* No prior treatment for esophageal cancer (surgery, laser, chemo- or radiotherapy)
* Oesophageal dilatation is allowed before or during the treatment, but prior esophageal prosthesis is not allowed
* Peripheral neuropathy <= NCI-CTC grade 1
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) <= 2
* Sufficient (oral or with gastrostomy) calorific intake (> 1000 Kcal/m2/day)
* Life expectancy >= 3 months
* Adequate bone marrow reserve, normal renal and liver functions:

  * Neutrophil count >= 1500/mm³
  * Platelet count >= 100,000/mm³
  * Hemoglobin >= 10 g/dl (after transfusion, if necessary)
  * Creatinine levels <= 1.5 x the upper normal limit of institutional values (ULN)
  * Total bilirubin level < 1.5 x ULN
  * ALT/AST < 2.5 x ULN
  * Prothrombin time >= 60%
* Laboratory values obtained the week preceding study entry
* Signed informed consent (prior to all study procedures)
* Start of treatment within 28 days of inclusion.

Exclusion Criteria:

* Metastatic disease except for third upper or cervical esophagus tumor with regional nodes, or third lower esophagus tumor with celiac nodes (M1a)
* Multiple carcinomas of the esophagus
* Small cell or undifferentiated carcinoma of the esophagus
* Complete dysphagia (grade 4 NCI-CTC); patient with exclusive parenteral nutrition.
* Weight loss > 20% normal body weight
* Pregnant or breast-feeding women
* Fertile patient not using adequate contraception
* Peripheral sensitive neuropathy with functional impairment
* Auditory disorders
* History of prior malignancies (other than cured non melanoma skin cancer, cured cervical carcinoma in situ or stage I or II node negative head and neck cancer cured > 3 years ago)
* Prior cervical, thoracic and abdominal radiotherapy with field overlapping the proposed oesophageal radiotherapy field
* Tracheo-oesophageal fistula or invasion of the tracheo-bronchial tree
* Previous myocardial infarction (inferior or equal to 6 months). Patients with a previous myocardial infarction superior to 6 months, could be included only if: no transient ischemia is shown by thallium myocardial scintigraphy and favourable advice for chemotherapy is obtained from a cardiologist.
* Other serious illness or medical conditions (such as symptomatic coronary disease, left ventricular failure or uncontrolled infection)
* Arterial disease stage II to IV according to the Leriche and Fontaine classification
* Treatment with any other experimental drugs or participation in another clinical trial within 30 days of study screening
* Concurrent treatment with any other anti-cancer therapy
* Concurrent treatment with phenytoin and yellow fever vaccine; geographical, social or psychological circumstances preventing regular follow-up.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients having completed the full treatment and Endoscopic complete response rate | at the end of the study

SECONDARY OUTCOMES:
Toxicity profile (NCI-CTC). | evaluated each week

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France